CLINICAL TRIAL: NCT01666886
Title: Efficacy of Additional Titration During Oral Appliance Treatment for Sleep-disordered Breathing.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Principal Investigator, ethisch.comite@uza.be, Ethics Committee Antwerp Univerity Hospital, University Hospital, Antwerp
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: EC 12/30/243
Record Dates: First submitted 2012-08-14; First posted 2012-08-16 (Estimated); Last update posted 2021-01-20 (Actual); Status verified 2021-01

CONDITIONS: Obstructive Sleep Apnea Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Occlusal Splints

ARMS (1):
- Mandibular Advancement Device (MAD) (Experimental): Mandibular advancement during therapy with a mandibular advancement device (MAD) in 90% of maximal protrusion
  Interventions: Device: Mandibular Advancement Device (MAD)

INTERVENTIONS:
Device: Mandibular Advancement Device (MAD)

SUMMARY:
In the protocol "Predicting therapeutic outcome of mandibular advancement device treatment in obstructive sleep apnea (PROMAD)", 100 patients with obstructive sleep apnea are included and started MAD treatment at 75% of maximal protrusion. All patients underwent polysomnography with MAD in situ to evaluate the effect of the MAD on severity of sleep apnea. If the results of the polysomnography with MAD are unsuccessful (defined as a reduction in AHI with the MAD in situ of less than 50% compared to baseline), the therapy needs to be adjusted. Finding the most effective protrusion should be a weighted compromise between efficacy and side-effects of MAD therapy.

In patients with insufficient results on the polysomnography with the MAD at 75% of maximal protrusion, the MAD will be further adjusted until 90% of the maximal protrusion measured at the follow-up visit after the polysomnography with the MAD. After habituation and adaptation period but within 2 months after the first polysomnography with MAD, a new polysomnography will be performed to assess the effect of the 90% protruded position.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Body Mass Index (BMI) ≤ 35 kg/m²
* OSAS, as defined by the American Academy of Sleep Medicine Task Force
* apnea-hypopnea index (AHI) < 50
* incomplete elimination of apneas and/or hypopnea during therapy with mandibular advancement device in 75% of maximal protrusion

Exclusion Criteria:

* Other sleep disorders (i.e. parasomnias)
* Invasive upper airway surgery for sleep-disordered breathing
* Known genetic disorders with craniofacial and/or upper airway malformations
* Use of benzodiazepine and/or antidepressants
* Known history of psychiatric disease
* Known history of fibromyalgia and/or chronic fatigue syndrome
* Dental contra-indications: functional restrictions of the temporomandibular joint, insufficient dentition with pathological changes, insufficient retention for MAD use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2012-08 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Polysomnographic efficacy | 3 to 6 months after start of therapy
  Polysomnographic re-evaluation of the severity of sleep apnea (apnea/hypopnea index).

CONTACTS AND LOCATIONS:
Locations (1):
- Antwerp University Hospital, Wilrijk, Antwerp, Belgium